CLINICAL TRIAL: NCT05525481
Title: Predicting an Accurate Tamoxifen Dose: a Feasibility Study in Patients With Hormone Sensitive Breast Cancer
Brief Title: Tamoxifen Prediction Study in Patients With ER+ Breast Cancer
Acronym: PREDICTAM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S. L. W. (Stijn) Koolen, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81896.078.22
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: ER+ Breast Cancer
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Non-randomized, single-center, single-arm, MIPD intervention study
Masking Description: One blood sample will be taken blindly and will be measured after the end of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): This is a single-arm trial. We only have one experimental arm. The control arm will be provided by another study.
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Hormone therapy

SUMMARY:
Adjuvant treatment with tamoxifen is the standard of care for women with estrogen receptor positive (ER+) breast cancer. Tamoxifen is converted to endoxifen, its active metabolite, via CYP2D6 enzymes. The literature states that an endoxifen concentration of at least 16 nmol/L is needed to produce a therapeutic effect (4). Therapeutic Drug Monitoring (TDM) has been proven to be a successful technique to reach the 16 nmol/L endoxifen threshold after 6 months. However, in general TDM can only be used when a drug is in steady-state, which for endoxifen is reached after 3 months for normal metabolizers. For poor- and intermediate metabolizers, the time until steady-state is presumably even longer. This could possibly result in undertreatment within the first 3 to 6 months of tamoxifen treatment. In this study, model-informed precision dosing (MIPD) will be used to counter this problem. The Pharmacokinetic-model, which is used for MIPD, includes CYP2D6 genotype, co-medication, age, body height, BMI and CYP2D6/CYP3A inhibitor use to predict a patient tailored dose. Using MIPD, our aim is to decrease the proportion of patients that are undertreated within the first three months of tamoxifen treatment.

DETAILED DESCRIPTION:
Tamoxifen, a selective estrogen receptor modulator, is currently the standard-of-care adjuvant treatment of breast cancer. Tamoxifen is a prodrug and particularly exerts its effect through its most active metabolite endoxifen. Cytochrome P450 (CYP) enzymes, in particular CYP2D6, convert tamoxifen to endoxifen. Polymorphisms in the CYP2D6 gene can hamper CYP2D6 activity and subsequently lead to decreased concentrations of endoxifen. Madlensky et al. found a direct association between endoxifen concentrations and breast cancer recurrence in a retrospective cohort. Patients with endoxifen concentrations below 16 nmol/L had a 30% higher risk of breast cancer recurrence than patients with endoxifen concentrations above this threshold. Madlensky et al. also found that CYP2D6 intermediate- and poor metabolizer phenotypes were associated with endoxifen levels below the 16 nmol/L threshold. The association between CYP2D6 phenotypes and endoxifen levels has since been confirmed by several other studies. In several retrospective studies, approximately 20-24% of tamoxifen patients do not reach the 16 nmol/L endoxifen threshold at steady state. Therapeutic drug monitoring (TDM) could be used to increase the probability of reaching this threshold to 89% after 6 months. With TDM, the dose is corrected after reaching steady state and patients are often only adequately treated after 3 to 6 months. To counter this problem and predict the correct tamoxifen dose at baseline, model-informed precision dosing (MIPD) could be used. In prior research at the Erasmus MC a population-pharmacokinetic (POP-PK) model has been developed. POP-PK-modeling is a mathematical modeling technique that describes the pharmacokinetics of a drug for each individual based on patient characteristics. A POPPK model can describe and predict the absorption, distribution, metabolism and elimination of a drug in the body and predict blood concentration-time profiles prior to actual administration of the drug. In previous, not yet published research we have developed a POP-PK model to describe tamoxifen and endoxifen pharmacokinetics. In this model we have evaluated the activity of different single nucleotide polymorphisms (SNP's) on a continuous scale. In addition the concomitant administration of CYP3A4 and CYP2D6 inhibitors influenced endoxifen formation. Whereas age significantly influenced tamoxifen clearance, BMI and height affected the endoxifen formation rate and tamoxifen clearance respectively.

After careful retrospective validation the validity of our model can be tested by prospectively predicting the best dose for each patient. Using Monte-Carlo simulations we estimated that when using the standard dose of 20 mg tamoxifen, 23% of all patients will not reach endoxifen steady-state concentration >16 nM. Using model-informed precision dosing, the proportion of patients that reach steady-state endoxifen concentrations above 16 nmol/L will be 91%. Out of these final 9%, 66% of all patients will not reach 16 nM using the highest registered dose of 40 mg. If the POP-PK model could adequately identify this patient group, that will not reach the 16 nM threshold with the highest prescribed dose of 40 mg, they could in the future be treated differently from the start of adjuvant therapy. An example of this are aromatase inhibitors.

The primary aim of this study is to increase the proportion of patients that reach an endoxifen level of 16 nM after reaching steady state endoxifen plasma concentrations using MIPD. In this study we will be prospectively validating a POP-PK model and evaluate the feasibility of MIPD for routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. WHO Performance Status ≤ 1 (see Appendix A);
3. Patients with primary breast cancer, with a prescription for adjuvant tamoxifen treatment;
4. Willing to abstain from strong and moderate CYP3A4 or CYP2D6 inhibitors or inducers, according to: CYTOCHROME P450 DRUG INTERACTION TABLE - Drug Interactions (iu.edu);
5. Able and willing to sign the Informed Consent Form;
6. Able and willing to undergo blood sampling for PK analysis.

Exclusion Criteria:

1. Patients with known alcoholism, drug addiction and/or psychiatric or physiological condition which in the opinion of the investigator would impair treatment compliance;
2. > 2 weeks of tamoxifen treatment before inclusion;
3. Patients who's endoxifen levels have been used for therapeutic drug monitoring in the past.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females.
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | Begin-end (3 months)
  The primary endpoint is the proportion of patients who reach an endoxifen level of 16 nmol/L or higher.

SECONDARY OUTCOMES:
Secondary outcome 1 | Begin-end (3 months)
  The total success rate (> 16 nmol/L and < 32 nmol/L) of the POP-PK model as well as in different groups, stratified by dosage as predicted by the POP-PK model.
Secondary outcome 2 | Begin-end (3 months)
  The predictive value of the POP-PK model for patients who do not reach the 16 nmol/L endoxifen threshold with the highest prescribed tamoxifen dose of 40 mg.
Secondary outcome 3 | Begin-end (3 months)
  The correlation between the endoxifen values from an early blood sample (4-6 weeks after start of treatment) and the steady-state concentration of endoxifen.
Secondary outcome 4 | Begin-end (3 months)
  The difference in incidence of side-effects and quality of life between baseline and 3 months after tamoxifen treatment as determined by FACT-ES questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands